CLINICAL TRIAL: NCT03648268
Title: Network Mediation of Experiential and Expressive Deficits in Psychotic Disorders
Brief Title: Using Transcranial Magnetic Stimulation (TMS) to Understand 'Negative' Symptoms of Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Mclean Hospital (Other); Harvard University (Other)
Responsible Party: Principal Investigator, Roscoe Brady, Assistant Professor of Psychiatry, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2018P000321
Record Dates: First submitted 2018-08-21; First posted 2018-08-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Schizophrenia; Negative Type; Schizophrenic; Schizo Affective Disorder
Keywords: brain; networks; schizophrenia
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: There will be four groups: an active DLPFC TMS group, an active TMS cerebellum group, a sham DLPFC group, and a sham cerebellum group. Participants will be randomized to one of these group groups, and they will receive that type of stimulation for the entire study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The subjects, care providers, investigators and outcome assessors will all be blinded as to the randomization sequence, and thus will be blinded as to sham vs active TMS status. Blinding codes are used to determine which side of an active/passive Magpro coil (cool B65 A/P, Magventure A/S, Denmark) is used for stimulation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Active DLPFC rTMS (Active Comparator): Active repetitive Transcranial Magnetic Stimulation (rTMS) with iTBS pattern to the right DLPFC at 80% of active motor threshold.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation (rTMS)
- Sham DLPFC rTMS (Sham Comparator): Sham repetitive Transcranial Magnetic Stimulation (rTMS) with iTBS pattern to the right DLPFC
  Interventions: Device: repetitive Transcranial Magnetic Stimulation (rTMS)
- Active cerebellum rTMS (Active Comparator): Active repetitive Transcranial Magnetic Stimulation (rTMS) with iTBS pattern to the cerebellum at 100% of active motor threshold.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation (rTMS)
- Sham cerebellum rTMS (Sham Comparator): Sham repetitive Transcranial Magnetic Stimulation (rTMS) with iTBS pattern to the cerebellum
  Interventions: Device: repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation (rTMS) — rTMS is a technique of TMS that allows the selective external manipulation of neural activity in a non-invasive manner. During TMS, a rapidly changing current is passed through an insulated coil placed against the scalp. This generates a temporary magnetic field that in turn induces electrical current in neurons and allows the modulation of neural circuitry. The combination of TMS with fMRI allows the selective targeting and modulation of brain networks. The repeated application of rTMS can cause long term changes in behavior and task performance that is reflected in altered brain network connectivity.
  The pattern of rTMS will consist of either:
  intermittent Theta Burst Stimulation (iTBS) pattern consisting of 2 s trains of 3 pulses at 50 Hz, repeated at 5 Hz, every 10s for a total of 600 pulses.
  OR
  sham stimulation
  Other Names: iTBS

SUMMARY:
The main purpose of this study is to learn how transcranial magnetic stimulation (TMS) helps improve negative symptoms of schizophrenia. These 'negative symptoms' include anhedonia (the inability to enjoy things), low motivation, and decreased facial expression.

TMS is a noninvasive way of stimulating the brain. TMS uses a magnetic field to cause changes in activity in the brain. The magnetic field is produced by a coil that is held next to the scalp. In this study we will be stimulating the brain to learn more about how TMS may improve these symptoms from schizophrenia.

DETAILED DESCRIPTION:
This study proposes to test the hypothesis that the medication refractory experiential (anhedonia and amotivation) and expressive deficits named 'negative symptoms' are mediated by network pathophysiology and the functional connectivity of a cerebellar-prefrontal cortical network mediates the severity of these deficits. To accomplish this participants will be recruited who are diagnosed with schizophrenia or schizoaffective disorder who demonstrate negative symptoms despite stable outpatient treatment.

Participants will undergo an initial screening session to complete informed consent and undergo baseline assessments of negative symptom severity. These assessments include reporter-based measures such as the Positive And Negative Syndrome Scale (PANSS) as well as quantitative tests of amotivation/anhedonia and diminished expressivity.

Participants will then undergo an MRI scan that includes structural and resting state functional magnetic resonance imaging (rsfMRI). These rsfMRI images will be used to isolate individual resting-state networks for targeting of rTMS modulation.

Participants will then undergo five days of twice daily rTMS sessions in one of the four arms of this study.

One week after the last rTMS session, Participants will undergo follow-up MRI imaging and the same assessments described above.

Aims:

Aim 1: To determine if network dysconnectivity is causally linked to negative symptom severity and if amelioration of this dysconnectivity results in reduced symptom severity. Symptom severity will be measured via both reporter-based and quantitative measures.

Aim 2: To determine if the relationship between functional connectivity and symptom severity arises from interactions between specific nodes of the default mode network (DMN): the cerebellum and DLPFC, or is the result of interactions between multiple nodes in the DMN (both cerebral and cerebellar).

Exploratory Aim: As an exploratory aim, additional genetic data will be collected which may be related to TMS efficacy. Hypothesis: Brain-derived neurotrophic factor (BDNF) homozygous val-allele carriers of the val66met BDNF gene will show greater response than met-carriers.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-55 years
* At pre-visit screening (see attached phone screening questionnaire): participants must report that they have been given a diagnosis of schizophrenia or schizoaffective disorder by a mental health professional
* Must be able to read, speak, and understand English
* Must be judged by study staff to be capable of completing the study procedures
* Diagnosis of schizophrenia or schizoaffective disorder according to DSM-V criteria and confirmed by SCID
* Participants will be in stable outpatient treatment with no recent (within the past 30 days) hospitalizations or changes in their mediation regimens

Exclusion Criteria:

* DSM-V intellectual disability
* substance use disorder within the past three months
* Ambidexterity (the EEfRT task assumes participants are not ambidextrous)
* Any history of progressive or genetic neurological disorder (e.g. Parkinson's disease, multiple sclerosis, tubular sclerosis, Alzheimer's Disease) or acquired neurological disease (e.g. stroke, traumatic brain injury, tumor), including intracranial lesions
* History of head trauma resulting in any loss of consciousness (>15 minutes) or neurological sequelae
* Current history of poorly controlled headaches including chronic medication for migraine prevention
* History of fainting spells of unknown or undetermined etiology that might constitute seizures
* History of seizures, diagnosis of epilepsy, or immediate (1st degree relative) family history epilepsy with the exception of a single seizure of benign etiology (e.g. febrile seizures) in the judgment of a board-certified neurologist
* Chronic (particularly) uncontrolled medical conditions that may cause a medical emergency in case of a provoked seizure (cardiac malformation, cardiac dysrhythmia, asthma, etc.)
* Any metal in the brain or skull (excluding dental fillings) or elsewhere in the body unless cleared by the responsible covering MD (e.g. MRI compatible joint replacement)
* Any devices such as pacemaker, medication pump, nerve stimulator, TENS unit, ventriculo-peritoneal shunt unless cleared by the responsible covering MD
* All female participants of child bearing age will be required to have a pregnancy test; any participant who is pregnant will not be enrolled in the study
* Medications will be reviewed by the responsible covering physician and a decision about inclusion will be made based on the participant's past medical history, drug dose, history of recent medication changes or duration of treatment, and use of CNS active drugs. The published TMS guidelines review of medications to be considered with rTMS will be taken into consideration given their described effects on cortical excitability measures.
* Any changes in medications or hospitalizations within the past 30 days.
* Subjects who, in the investigator's opinion, might not be suitable for the study or would be unable to tolerate the study visit

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Change in Negative Symptom Severity | Before treatment (Baseline) and 1 week post treatment
  We will evaluate the effect of sham vs active rTMS on negative symptom severity in the group with Cerebellar targeted rTMS and in the group with DLPFC targeted rTMS

SECONDARY OUTCOMES:
Change in Cerebellar - Prefrontal Functional Connectivity | Before treatment (Baseline) and 1 week post treatment
  We will evaluate the effect of sham vs active rTMS on cerebellar-prefrontal cortex functional connectivity in the group with Cerebellar targeted rTMS and in the group with DLPFC targeted rTMS
Change in Auditory Hallucination Severity | Before treatment (Baseline) and 1 week post treatment
  We will evaluate the effect of sham vs active rTMS on the frequency and severity of auditory hallucinations in the group with Cerebellar targeted rTMS and in the group with DLPFC targeted rTMS

CONTACTS AND LOCATIONS:
Overall Officials: Roscoe Brady, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
This study will adhere to the published Data Sharing Expectations for NIMH-funded Clinical Trials outlined in NOT-MH-14-015. We will share data collected in these experiments with the National Database for Clinical Trials related to Mental Illness using its GUID and Data Dictionary technology.

REFERENCES:
- [Background] Rabinowitz J, Levine SZ, Garibaldi G, Bugarski-Kirola D, Berardo CG, Kapur S. Negative symptoms have greater impact on functioning than positive symptoms in schizophrenia: analysis of CATIE data. Schizophr Res. 2012 May;137(1-3):147-50. doi: 10.1016/j.schres.2012.01.015. Epub 2012 Feb 6. PMID 22316568
- [Background] Robertson BR, Prestia D, Twamley EW, Patterson TL, Bowie CR, Harvey PD. Social competence versus negative symptoms as predictors of real world social functioning in schizophrenia. Schizophr Res. 2014 Dec;160(1-3):136-41. doi: 10.1016/j.schres.2014.10.037. Epub 2014 Nov 7. PMID 25468184
- [Background] Roth BJ, Cohen LG, Hallett M. The electric field induced during magnetic stimulation. Electroencephalogr Clin Neurophysiol Suppl. 1991;43:268-78. PMID 1773764
- [Background] Roth BJ, Saypol JM, Hallett M, Cohen LG. A theoretical calculation of the electric field induced in the cortex during magnetic stimulation. Electroencephalogr Clin Neurophysiol. 1991 Feb;81(1):47-56. doi: 10.1016/0168-5597(91)90103-5. PMID 1705219
- [Background] Walsh V, Cowey A. Transcranial magnetic stimulation and cognitive neuroscience. Nat Rev Neurosci. 2000 Oct;1(1):73-9. doi: 10.1038/35036239. PMID 11252771
- [Background] Eldaief MC, Halko MA, Buckner RL, Pascual-Leone A. Transcranial magnetic stimulation modulates the brain's intrinsic activity in a frequency-dependent manner. Proc Natl Acad Sci U S A. 2011 Dec 27;108(52):21229-34. doi: 10.1073/pnas.1113103109. Epub 2011 Dec 12. PMID 22160708
- [Background] Yeo BT, Krienen FM, Sepulcre J, Sabuncu MR, Lashkari D, Hollinshead M, Roffman JL, Smoller JW, Zollei L, Polimeni JR, Fischl B, Liu H, Buckner RL. The organization of the human cerebral cortex estimated by intrinsic functional connectivity. J Neurophysiol. 2011 Sep;106(3):1125-65. doi: 10.1152/jn.00338.2011. Epub 2011 Jun 8. PMID 21653723
- [Background] Power JD, Cohen AL, Nelson SM, Wig GS, Barnes KA, Church JA, Vogel AC, Laumann TO, Miezin FM, Schlaggar BL, Petersen SE. Functional network organization of the human brain. Neuron. 2011 Nov 17;72(4):665-78. doi: 10.1016/j.neuron.2011.09.006. PMID 22099467
- [Background] Demirtas-Tatlidede A, Freitas C, Cromer JR, Safar L, Ongur D, Stone WS, Seidman LJ, Schmahmann JD, Pascual-Leone A. Safety and proof of principle study of cerebellar vermal theta burst stimulation in refractory schizophrenia. Schizophr Res. 2010 Dec;124(1-3):91-100. doi: 10.1016/j.schres.2010.08.015. PMID 20817483
- [Background] Garg S, Sinha VK, Tikka SK, Mishra P, Goyal N. The efficacy of cerebellar vermal deep high frequency (theta range) repetitive transcranial magnetic stimulation (rTMS) in schizophrenia: A randomized rater blind-sham controlled study. Psychiatry Res. 2016 Sep 30;243:413-20. doi: 10.1016/j.psychres.2016.07.023. Epub 2016 Jul 16. PMID 27450744
- [Background] Schmahmann JD. An emerging concept. The cerebellar contribution to higher function. Arch Neurol. 1991 Nov;48(11):1178-87. doi: 10.1001/archneur.1991.00530230086029. PMID 1953406
- [Background] Schmahmann JD. Dysmetria of thought: clinical consequences of cerebellar dysfunction on cognition and affect. Trends Cogn Sci. 1998 Sep 1;2(9):362-71. doi: 10.1016/s1364-6613(98)01218-2. PMID 21227233
- [Background] Andreasen NC, Paradiso S, O'Leary DS. "Cognitive dysmetria" as an integrative theory of schizophrenia: a dysfunction in cortical-subcortical-cerebellar circuitry? Schizophr Bull. 1998;24(2):203-18. doi: 10.1093/oxfordjournals.schbul.a033321. PMID 9613621
- [Background] Parker KL, Narayanan NS, Andreasen NC. The therapeutic potential of the cerebellum in schizophrenia. Front Syst Neurosci. 2014 Sep 15;8:163. doi: 10.3389/fnsys.2014.00163. eCollection 2014. PMID 25309350
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552